CLINICAL TRIAL: NCT07257757
Title: Evaluation of the Analgesic Efficacy of Fascia Iliaca Compartment Block in Patients Undergoing Total Knee Arthroplasty With Intra-Articular Injection: a Retrospective Cohort Study
Brief Title: Fascia Iliaca Compartment Block in Total Knee Arthroplasty With Intra-Articular Injection
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Zafer Gün, Research Assistant, Kırıkkale University
Other Study IDs: KirikkaleU-2024.06.01
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Total Knee Arthroplasty (Postoperative Pain)
Keywords: Postoperative; Patient Satisfaction; Pain; Bleeding; Peripheral Nerve Block; Continuous Fascia Iliaca Comparment Block; Intra-articular Injection
MeSH Terms: conditions — Pain, Postoperative; Patient Satisfaction; Pain; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Total knee arthroplasty cases where only intra-articular injection was performed
- Continuous Fascia Iliaca Compartment Block Group: Total knee arthroplasty cases in which continuous fascia iliaca compartment block is performed in addition to intra-articular injection

SUMMARY:
The purpose of our study is to retrospectively investigate the effect of continuous fascia iliaca compartment block in total knee arthroplasty cases in addition to intraoperative intra-articular injection.

DETAILED DESCRIPTION:
Postoperative pain management is of great importance in orthopedic surgeries. Inadequate analgesia following total knee arthroplasty increases the risk of side effects such as thromboembolism, myocardial ischemia, pulmonary dysfunction, paralytic ileus, urinary retention, and postoperative bleeding, thereby prolonging hospital stays.

Recently, fascia iliaca compartment block (FICB) has been frequently used to treat pain following knee replacement surgery. However, there are only a limited number of studies demonstrating the effectiveness of this method for postoperative analgesia. Sensory innervation of the lower extremity is primarily provided by four main nerves and their branches. These are the sciatic nerve, femoral nerve, obturator nerve, and lateral femoral cutaneous nerve. FICB is a compartment block in which local anesthetic is injected under the iliac fascia to block the femoral nerve, obturator nerve, and lateral femoral cutaneous nerve. The iliac fascia is the second fascial plane encountered when examining the proximal lower extremity with ultrasound (USG), extending immediately beneath the fascia latae. The goal is to place the needle tip under the iliac fascia, a few centimeters away from the femoral artery. Then, a single dose of local anesthetic can be administered under the iliac fascia, or a catheter can be placed in this area with ultrasound guidance.

Cocktails containing local anesthetic, narcotic analgesic, epinephrine, methylprednisolone, and cefuroxime are injected periarticularly for the preemptive treatment of pain following knee replacement surgery. This method, one of the multimodal protocols, is used to minimize the use of parenteral narcotics in order to protect against side effects.

Regional blocks are simple techniques that not only improve postoperative pain control but also reduce postoperative opioid requirements, shorten hospital stays, increase patient satisfaction, and lead to better clinical outcomes after total knee arthroplasty.

In our clinic, continuous fascia iliaca compartment block is applied for postoperative analgesia in total knee arthroplasty cases. The aim of this study is to retrospectively investigate the effect of continuous fascia iliaca compartment block in addition to intraoperative intra-articular injection on postoperative analgesia, postoperative bleeding and patient satisfaction in total knee arthroplasty cases.

ELIGIBILITY:
Inclusion Criteria:

* Total knee arthroplasty cases with or without continuous fascia iliaca compartment block
* Patients with ASA criteria 1-2-3

Exclusion Criteria:

* Patients whose records cannot be accessed
* Patients with ASA criteria 4-5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent unilateral total knee arthroplasty at the Orthopedics and Traumatology Clinic of Kırıkkale University Faculty of Medicine Hospital and received postoperative analgesia using different methods
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Postoperative 24 hours
  The visual analog scale is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
Rating levels of satisfaction | Posoperative 24 hours
  A possible scale is then: "Not at all Satisfied," "Partly Satisfied," "Satisfied," "More than Satisfied," "Very Satisfied," numbering 1 to 5 as an interval scale.
Recording of surgical drain output | Postoperative 24 hours
  Monitoring the output from surgical drains is important part of post-operative care. It is a measurement method that allows us to monitor the amount of bleeding in a patient after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Kevser PEKER, Assoc. Prof., Study Director — Kırıkkale University
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)